CLINICAL TRIAL: NCT00553384
Title: Physiological Effects of Androstadienone Exposure
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: LVO-0619
Record Dates: First submitted 2007-11-01; First posted 2007-11-05 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: smell; olfaction; androstadienone; women; pheromones; Healthy Volunteers; Physiological Effects of Androstadienone Exposure
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The reason for doing this research is to understand why different people show different responses when they smell an odor called androstadienone. Androstadienone is a chemical found in male sweat. Other studies have shown that smelling this chemical can cause people to experience sweating, changes in skin temperature, and changes in a stress hormone call cortisol. These responses, which are called "physiological effects," are stronger in some people than in others.

We are interested in finding out whether these individual differences are genetic, that is caused by differences in our genes. Humans have about 1000 genes for odorant receptors. These are the molecules that bind and detect odor molecules in our nose and allow us to respond to so many different odors. It has been shown that some of these genes exist in two forms: a functional one and one that has been mutated and is therefore no longer functional.

We think that people who do not respond to a specific odor may carry the non-functional form of the gene for the receptor that detects the odor molecule. To test this idea we want to find people who respond strongly to a specific smell, and compare their odorant receptor genes with those of people who respond weakly to the odor.

DETAILED DESCRIPTION:
The study consists of five visits. The first visit is a screening visit at which the eligibility of the subject is determined and a blood sample is taken. At this visit, the subject is also given ovulation test strips and instructions to perform urine-based ovulation self-tests at home for a period of several days following the onset of menstruation. The subject is instructed to test her urine at home until an LH surge is detected.

When the subject ovulates and is available for a visit she will come to the Rockefeller University Hospital within one day of detecting an LH surge for the first of four Test Sessions.

The four Test Sessions are identical with the exception that the subject is exposed to a different odor stimulus.

We will be measuring:

1. skin temperature
2. sweating, as measured by skin conductance
3. salivary cortisol levels.
4. mood

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult women between 18-35 years of age.
* Only subjects whose threshold to either vanillin or isovaleric acid is in the 90th percentile of the population tested in LVO-0539-0507 and who do not report any clinical conditions that may disturb their sense of smell will be enrolled in the study.

Exclusion Criteria:

* Use of oral contraceptives over the last 3 months
* Pregnancy
* Allergies to odors or fragrances
* History of nasal illness
* Irregular menstrual periods
* History of medical conditions that reduced or abolished sense of smell, such as: head injury, cancer therapy, radiation to the head and neck, or alcoholism.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult women between 18-35 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2007-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Skin temperature, skin conductance and salivary cortisol level. | Monthly over approximately a 5 month period/volunteer

SECONDARY OUTCOMES:
The ability to detect odor. | Monthly over a 5 month period.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Vosshall, Ph.D., Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University Hospital, New York, New York, United States